CLINICAL TRIAL: NCT04517162
Title: Effect of Collagen-Polyvinylpyrrolidone for the Treatment of Hyperinflammation and the Pulmonary Fibrosis in COVID-19 Patients. Double Blind Placebo-controlled Pilot Trial
Brief Title: Intramuscular Effect of Polymerized Type I Collagen on the Cytokine Storm in COVID-19 Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Janette Furuzawa Carballeda (Other)
Responsible Party: Sponsor-Investigator, Janette Furuzawa Carballeda, Medical science resercher, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRE-3412-20-21-1
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Cytokine Storm; Regulation of Inflammatory Response; Pulmonary Fibrosis
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Pulmonary Fibrosis | interventions — collagen-PVP

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo-controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator or polymerized type I collagen (Active Comparator): 1.5 mL of polymerized type I collagen every 12 h for 3 days and then every 24 h for 4 days (in total 10 injections in 7 days)
  Interventions: Drug: Collagen-Polyvinylpyrrolidone
- Placebo comparator o placebo (Placebo Comparator): 1.5 mL of placebo, every 12 h for 3 days and then every 24 h for 4 days (in total 10 injections in 7 days)
  Interventions: Drug: Collagen-Polyvinylpyrrolidone

INTERVENTIONS:
Drug: Collagen-Polyvinylpyrrolidone — 1.5 mL of polymerized-type I collagen or placebo, every 12 h for 3 days and then every 24 h for 4 days (in total 10 injections in 7 days)
  Other Names: Fibroquel; Polymerized-Type I Collagen; polymerized type I collagen

SUMMARY:
SARS-CoV-2 infection induces a hyperinflammatory syndrome, causing the acute respiratory distress syndrome, massive lung cell destruction and, as a plausible sequelae, pulmonary fibrosis in COVID-19 patients.

Current focus has been on the development of novel immunosuppressant therapies, in order to control the cytokine storm in COVID-19 patients. Thus, the effect of steroids, intravenous immunoglobulin, non-steroidal immunosuppressants, selective cytokine blockade, JAK/STAT pathway inbhibition, and mesenchymal precursor cells have been evaluated. Based on the above information, we propose COLLAGEN-POLYVINYLPYRROLIDONE (Distinctive name: FibroquelMR, active substance: Collagen-polyvinylpyrrolidone, pharmaceutical form: intramuscular injectable solution, with sanitary registration No. 201M95 SSA IV and SSA code: 010 000 3999) as a potential drug for the downregulation of the cytokine storm. Polymerized type I collagen reduces the expression of IL-1β, IL-8, TNF-alpha, TGF-β1, IL-17, Cox-1, leukocyte adhesion molecules (ELAM-1, VCAM- 1 and ICAM-1), some other mediators of inflammation and increases the levels of IL-10 and the number of regulatory T cells. In addition, it promotes the mechanisms of inhibition of tissue fibrosis, without adverse effects in rheumatoid arthritis and osteoarthritis.

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo-controlled, randomized clinical trial that compares PTIC with placebo in adult outpatients with confirmed COVID-19. The study was approved by the institutional review board at Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ, reference no. IRE 3412-20-21-1) and was conducted in compliance with the Declaration of Helsinki (World Medical Association. World Medical Association Declaration of Helsinki. JAMA. 2013;310(20):2191-2194.), the Good Clinical Practice guidelines, and local regulatory requirements. All participants will provide written informed consent.

Trial candidates will be identified in a prospective database of patients that go to a medical appointment at the hospital and be discharged home with a diagnosis of COVID-19 and symptomatic treatment. Diagnosis will base on suggestive symptoms (fever, headache, cough or dyspnea, plus another symptom such as malaise, myalgias, arthralgias, rhinorrhea, throat pain, conjunctivitis, vomiting or diarrhea) and positive real-time reverse-transcription polymerase chain (RT-PCR).

Staff will reach candidates via telephone calls and inform them about the purpose of the study. Once in the hospital study site, and after verifying inclusion (suggestive symptoms and PCR) and exclusion criteria, patients will sign the informed consent before being randomly allocated to either PTIC or matching placebo. Exclusion criteria includes hypersensitivity to PTIC or any of its excipients, COVID-19 patients that require hospitalization, all pregnant or breast-feeding patients, patients with chronic kidney disease as determined by calculating an estimated glomerular filtration rate (eGFR), or need for hemodialysis or hemofiltration, decompensated cirrhosis, congestive heart failure (New York Heart Association class III or IV), patients with cerebrovascular disease, autoimmune disease, cancer, multiorgan failure or immunocompromised (solid organ transplant recipient or donor, bone marrow transplant recipient, AIDS, or taking immunosuppressant biologic drugs or corticosteroids).

During the first day of enrollment, candidates will receive the study supplies that consist of the study medication or placebo, a pulse oximeter, and a symptom questionnaire booklet. Patients will be instructed on how to administer the study medication, how to use the oxygen monitor and how to complete the questionnaires. Also, staff will administer the first dose of study medication or placebo on site.

Phone contact will make daily during the first 3 days of the trial to address participants' questions, address any medication-related issues, and encourage completion of questionnaires. Additional phone calls will be conducted on a case-by-case basis when participant's survey data indicated values outside of expected ranges. For participants that will have a worsening disease course (89% or lower while breathing ambient air), study staff will recommend to attend at emergency department. If the patient will require hospitalization and treatment with dexamethasone, then patient will be eliminated from the study. Patients will be evaluated by staff on day 8, 15 and 97 (1, 7 and 90 days after last dose of medication or placebo, respectively).

Participants The study will include non-hospitalized adults with COVID-19 whose symptoms start within the previous 7 days counted from the first dose of study medication. Individuals will ask to provide personal information (date of birth, type of job, educational level, previous contact with infected individuals, and date of symptom onset), preexisting conditions (systemic hypertension, diabetes mellitus, cardiovascular disease, cerebrovascular disease, hypertriglyceridemia, dyslipidemia) and symptoms.

Real-time reverse-transcription polymerase chain Naso/oropharyngeal swab samples will obtain and send in a universal transport medium for viruses. Nucleic acid extraction will do using the NucliSens easy-MAG system (bioMérieux, Boxtel, Netherlands). RT-PCR will carry out in the Applied Biosystems 7500 thermocycler (Applied Biosystems, Foster City, CA, USA) using primers and conditions described elsewhere; the cycle threshold value for positivity will 38 (Corman VM, 2020).

Study sample According to a study completed previously in Mexico City (Valencia CA, 2008), the mean oxygen saturation readings of a selected elderly sample without cardiopulmonary comorbidities was 95.3 ± 1.7%. Since a notorious drop in such readings was not to be expected (due to the non-severe nature of disease in our sample of outpatients), it was arbitrarily decided that a difference of 2 percentage points (beyond the preceding standard deviation cutoff points) between groups would be clinically significant in this pilot study. In this regard, total sample size assuming alpha=0.05 and power=0.80 was 32. However, to increase the power to detect meaningful differences in frequency of cough between groups (a potential indicator of lung disease), it was decided to include 45 patients per group (based on a baseline frequency of 60% (Wang DA, 2020) and a reduction of symptom frequency by half with the experimental intervention, keeping alpha and power values fixed).

Randomization Patients will be randomized in a 1:1 fashion to PTIC or matching placebo. Randomization schedules will prepare in Excel, which displayed randomization assignment to the laboratory manager, who will prepare the study materials, including the study drug or placebo. All outcome assessors, investigators, and research staff who will be in contact with participants will blind to participant treatment assignment.

Intervention Participants will receive an intramuscular dose of either PTIC (1.5 ml, equivalent to 12.5 mg of collagen) every 12 h for 3 days and then every 24 h for 4 days, or matching placebo. Only acetaminophen or acetylsalicylic acid will allow as concomitant therapy.

Data collection Personal data, contact and exposure history, clinical presentation, chest computed (CT) tomography, laboratory tests, previous treatment and outcome data will collect both prospectively and from inpatient medical records. Laboratory data collected from each patient from study days 1 (baseline), 8 (1-day post-treatment), 15 (7 days post-treatment) and 97 (90 days post-treatment) will include complete blood count, coagulation profile, serum biochemical tests (including renal and liver function tests, electrolytes, lactate dehydrogenase, D dimer and creatine kinase), serum ferritin, and biomarkers of infection, such as procalcitonin. Chest CT scans will be done in all patients at baseline.

ELIGIBILITY:
Inclusion Criteria:

* According to the sample size calculation (Cohen's d calculation, using a 50% decrease in IP-10 as the expected effect size), 90 COVID-19 patients will be recruited (symptoms: cough, expectoration, odynophagia, dyspnea with or without fever; radiographic findings by imaging study: inflammatory infiltrates), of both sexes, older than 18 years.
* Participants will be enrolled, even when they do not have a laboratory-confirmed SARS-CoV-2 infection as determined by a positive reverse transcription, polymerase-chain-reaction (RT-PCR) assay result. Patients will be included if they have progressive disease consistent with ongoing SARS-CoV -2 infection.
* Patients with laboratory predictors of mild to severe disease (D-dimer> 1000 ng/ml; total lymphocytes <800 cells/µl, creatine phosphokinase> 2 times upper limit of the normal range; elevated troponins and ferritin> 300 µg/L) will be included.
* Only those patients who are negative to the intradermal reaction of polymerized type I collagen (subcutaneous application of 0.2 ml of the drug on the forearm, evaluation at 24-48h) will be included.
* Patients with mild to severe disease, peripheral oxygen saturation (SpO2) <92% on room air, or requiring supplemental oxygen, or mechanical ventilation will be recruited. There will be no limit to the duration of symptoms prior to enrollment.
* Only those patients who are not participating in another protocol and who are not receiving biological therapy and whose standardized therapy is suggested will be included (AmoxiClav or ceftriaxone, or azithromycin, clarithromycin or doxycycline, ivermectin, low molecular weight anticoagulants, paracetamol).
* All patients who agree to participate in the protocol and from whom written informed consent is obtained will be included.

Exclusion Criteria:

* All patients positive for intradermal reaction to polymerized type I collagen (allergy to study producto) will be excluded.
* All pregnant or breast-feeding patients, patients with chronic kidney disease as determined by calculating an estimated glomerular filtration rate (eGFR), or need for hemodialysis or hemofiltration, patients with cerebrovascular disease, autoimmune disease, cancer, multiorgan failure or immunodeficiencies (HIV, transplant patients, hematological diseases, patients with chemotherapy) will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-19 (Estimated); Study Completion 2021-06-19 (Estimated)

PRIMARY OUTCOMES:
Clinical primary Outcome measure | 14 days
  It will be considered as primary outcome if the patients meet the first criterion, or 2 of the remaining 3:
  1. No oxygen required to maintain oxygen saturation more than 92%,
  2. Decrease in severity category from Table 1 by at least 1 level, or
  3. Reduction in the time of symptoms, by at least 30% compared to placebo and baseline, or
  4. recovery of at least 30% the number of lymphocytes compared to placebo and baseline.

SECONDARY OUTCOMES:
Immunological secondary outcome measure | 3 months
  It will be considered as secondary outcome if the patients meet the first criterion, or 2 of the remaining 3:
  1. significant decrease in serum IP-10 (at least 30% compared to placebo and baseline), since this chemokine is directly associated with the progression and severity of COVID-19,
  2. significant decrease in serum pro-inflammatory cytokines (TNF-a, IL-1β, IL-7, at least 30% compared to placebo and baseline),
  3. significant decrease in the percentage of circulating effector T cells (at least 30% compared to placebo and baseline), or
  4. significant improvement from computerized axial tomography at re-examination. This improvement is defined as: a decrease of at least 40% in parenchymal attenuation, the appearance of ground glass, nodular opacities, thickening of interlobular septa and / or thickening of bronchial walls.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ochoa-Hein, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Luis A Septien-Stute, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Janette Furuzawa-Carballeda, PhD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Gonzalo Torres-Villalobos, MD, PhD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Daniel Azamar-Llamas, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Diego F Hernández-Ramírez, PhD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Elizabeth Olivares-Martínez, PhD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Data will be provided based on requirement

REFERENCES:
- [Result] Channappanavar R, Fehr AR, Vijay R, Mack M, Zhao J, Meyerholz DK, Perlman S. Dysregulated Type I Interferon and Inflammatory Monocyte-Macrophage Responses Cause Lethal Pneumonia in SARS-CoV-Infected Mice. Cell Host Microbe. 2016 Feb 10;19(2):181-93. doi: 10.1016/j.chom.2016.01.007. PMID 26867177
- [Result] Elhai M, Avouac J, Allanore Y. Circulating lung biomarkers in idiopathic lung fibrosis and interstitial lung diseases associated with connective tissue diseases: Where do we stand? Semin Arthritis Rheum. 2020 Jun;50(3):480-491. doi: 10.1016/j.semarthrit.2020.01.006. Epub 2020 Jan 28. PMID 32089354
- [Result] Feldmann M, Maini RN, Woody JN, Holgate ST, Winter G, Rowland M, Richards D, Hussell T. Trials of anti-tumour necrosis factor therapy for COVID-19 are urgently needed. Lancet. 2020 May 2;395(10234):1407-1409. doi: 10.1016/S0140-6736(20)30858-8. Epub 2020 Apr 9. No abstract available. PMID 32278362
- [Result] Furuzawa-Carballeda J, Lima G, Llorente L, Nunez-Alvarez C, Ruiz-Ordaz BH, Echevarria-Zuno S, Hernandez-Cuevas V. Polymerized-type I collagen downregulates inflammation and improves clinical outcomes in patients with symptomatic knee osteoarthritis following arthroscopic lavage: a randomized, double-blind, and placebo-controlled clinical trial. ScientificWorldJournal. 2012;2012:342854. doi: 10.1100/2012/342854. Epub 2012 Apr 1. PMID 22545014
- [Result] Furuzawa-Carballeda J, Munoz-Chable OA, Barrios-Payan J, Hernandez-Pando R. Effect of polymerized-type I collagen in knee osteoarthritis. I. In vitro study. Eur J Clin Invest. 2009 Jul;39(7):591-7. doi: 10.1111/j.1365-2362.2009.02154.x. PMID 19453649
- [Result] Furuzawa-Carballeda J, Munoz-Chable OA, Macias-Hernandez SI, Agualimpia-Janning A. Effect of polymerized-type I collagen in knee osteoarthritis. II. In vivo study. Eur J Clin Invest. 2009 Jul;39(7):598-606. doi: 10.1111/j.1365-2362.2009.02144.x. Epub 2009 Apr 23. PMID 19397687
- [Result] Furuzawa-Carballeda J, Alcocer-Varela J, Diaz de Leon L. Collagen-PVP decreases collagen turnover in synovial tissue cultures from rheumatoid arthritis patients. Ann N Y Acad Sci. 1999 Jun 30;878:598-602. doi: 10.1111/j.1749-6632.1999.tb07738.x. No abstract available. PMID 10415784
- [Result] Furuzawa-Carballeda J, Cabral AR, Zapata-Zuniga M, Alcocer-Varela J. Subcutaneous administration of polymerized-type I collagen for the treatment of patients with rheumatoid arthritis. An open-label pilot trial. J Rheumatol. 2003 Feb;30(2):256-9. PMID 12563677
- [Result] Furuzawa-Carballeda J, Fenutria-Ausmequet R, Gil-Espinosa V, Lozano-Soto F, Teliz-Meneses MA, Romero-Trejo C, Alcocer-Varela J. Polymerized-type I collagen for the treatment of patients with rheumatoid arthritis. Effect of intramuscular administration in a double blind placebo-controlled clinical trial. Clin Exp Rheumatol. 2006 Sep-Oct;24(5):514-20. PMID 17181919
- [Result] Furuzawa-Carballeda J, Krotzsch E, Barile-Fabris L, Alcala M, Espinosa-Morales R. Subcutaneous administration of collagen-polyvinylpyrrolidone down regulates IL-1beta, TNF-alpha, TGF-beta1, ELAM-1 and VCAM-1 expression in scleroderma skin lesions. Clin Exp Dermatol. 2005 Jan;30(1):83-6. doi: 10.1111/j.1365-2230.2004.01691.x. PMID 15663512
- [Result] Furuzawa-Carballeda J, Macip-Rodriguez P, Galindo-Feria AS, Cruz-Robles D, Soto-Abraham V, Escobar-Hernandez S, Aguilar D, Alpizar-Rodriguez D, Ferez-Blando K, Llorente L. Polymerized-type I collagen induces upregulation of Foxp3-expressing CD4 regulatory T cells and downregulation of IL-17-producing CD4(+) T cells (Th17) cells in collagen-induced arthritis. Clin Dev Immunol. 2012;2012:618608. doi: 10.1155/2012/618608. Epub 2011 Oct 19. PMID 22028728
- [Result] Furuzawa-Carballeda J, Ortiz-Avalos M, Lima G, Jurado-Santa Cruz F, Llorente L. Subcutaneous administration of polymerized type I collagen downregulates interleukin (IL)-17A, IL-22 and transforming growth factor-beta1 expression, and increases Foxp3-expressing cells in localized scleroderma. Clin Exp Dermatol. 2012 Aug;37(6):599-609. doi: 10.1111/j.1365-2230.2012.04385.x. Epub 2012 Jun 25. PMID 22731679
- [Result] Furuzawa-Carballeda J, Rojas E, Valverde M, Castillo I, Diaz de Leon L, Krotzsch E. Cellular and humoral responses to collagen-polyvinylpyrrolidone administered during short and long periods in humans. Can J Physiol Pharmacol. 2003 Nov;81(11):1029-35. doi: 10.1139/y03-101. PMID 14719037
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Krotzsch-Gomez FE, Furuzawa-Carballeda J, Reyes-Marquez R, Quiroz-Hernandez E, Diaz de Leon L. Cytokine expression is downregulated by collagen-polyvinylpyrrolidone in hypertrophic scars. J Invest Dermatol. 1998 Nov;111(5):828-34. doi: 10.1046/j.1523-1747.1998.00329.x. PMID 9804346
- [Result] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Result] Liang W, Liang H, Ou L, Chen B, Chen A, Li C, Li Y, Guan W, Sang L, Lu J, Xu Y, Chen G, Guo H, Guo J, Chen Z, Zhao Y, Li S, Zhang N, Zhong N, He J; China Medical Treatment Expert Group for COVID-19. Development and Validation of a Clinical Risk Score to Predict the Occurrence of Critical Illness in Hospitalized Patients With COVID-19. JAMA Intern Med. 2020 Aug 1;180(8):1081-1089. doi: 10.1001/jamainternmed.2020.2033. PMID 32396163
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Moreno-Alvarez P, Sanchez-Guerrero E, Martinez-Cordero E, Hernandez-Pando R, Campos MG, Cetina L, Bazan-Perkins B. Aerosolized polymerized type I collagen reduces airway inflammation and remodelling in a guinea pig model of allergic asthma. Lung. 2010 Apr;188(2):97-105. doi: 10.1007/s00408-009-9202-2. Epub 2009 Dec 9. PMID 19998041
- [Result] Olmos-Zuniga JR, Hernandez-Jimenez C, Diaz-Martinez E, Jasso-Victoria R, Sotres-Vega A, Gaxiola-Gaxiola MO, Villalba-Caloca J, Baltazares-Lipp M, Santillan-Doherty P, Santibanez-Salgado JA. Wound healing modulators in a tracheoplasty canine model. J Invest Surg. 2007 Nov-Dec;20(6):333-8. doi: 10.1080/08941930701772140. PMID 18097874
- [Result] Olmos-Zuniga JR, Silva-Martinez M, Jasso-Victoria R, Baltazares-Lipp M, Hernandez-Jimenez C, Buendia-Roldan I, Jasso-Arenas J, Martinez-Salas A, Calyeca-Gomez J, Guzman-Cedillo AE, Gaxiola-Gaxiola M, Romero-Romero L. Effects of Pirfenidone and Collagen-Polyvinylpyrrolidone on Macroscopic and Microscopic Changes, TGF-beta1 Expression, and Collagen Deposition in an Experimental Model of Tracheal Wound Healing. Biomed Res Int. 2017;2017:6471071. doi: 10.1155/2017/6471071. Epub 2017 May 11. PMID 28584818
- [Result] Saeidi A, Zandi K, Cheok YY, Saeidi H, Wong WF, Lee CYQ, Cheong HC, Yong YK, Larsson M, Shankar EM. T-Cell Exhaustion in Chronic Infections: Reversing the State of Exhaustion and Reinvigorating Optimal Protective Immune Responses. Front Immunol. 2018 Nov 9;9:2569. doi: 10.3389/fimmu.2018.02569. eCollection 2018. PMID 30473697
- [Result] Stebbing J, Phelan A, Griffin I, Tucker C, Oechsle O, Smith D, Richardson P. COVID-19: combining antiviral and anti-inflammatory treatments. Lancet Infect Dis. 2020 Apr;20(4):400-402. doi: 10.1016/S1473-3099(20)30132-8. Epub 2020 Feb 27. No abstract available. PMID 32113509
- [Result] Sun L, Louie MC, Vannella KM, Wilke CA, LeVine AM, Moore BB, Shanley TP. New concepts of IL-10-induced lung fibrosis: fibrocyte recruitment and M2 activation in a CCL2/CCR2 axis. Am J Physiol Lung Cell Mol Physiol. 2011 Mar;300(3):L341-53. doi: 10.1152/ajplung.00122.2010. Epub 2010 Dec 3. PMID 21131395
- [Result] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Result] Yang Y, Shen C, Li J, Yuan J, Wei J, Huang F, Wang F, Li G, Li Y, Xing L, Peng L, Yang M, Cao M, Zheng H, Wu W, Zou R, Li D, Xu Z, Wang H, Zhang M, Zhang Z, Gao GF, Jiang C, Liu L, Liu Y. Plasma IP-10 and MCP-3 levels are highly associated with disease severity and predict the progression of COVID-19. J Allergy Clin Immunol. 2020 Jul;146(1):119-127.e4. doi: 10.1016/j.jaci.2020.04.027. Epub 2020 Apr 29. PMID 32360286
- [Result] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Result] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- [Result] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Result] Zheng HY, Zhang M, Yang CX, Zhang N, Wang XC, Yang XP, Dong XQ, Zheng YT. Elevated exhaustion levels and reduced functional diversity of T cells in peripheral blood may predict severe progression in COVID-19 patients. Cell Mol Immunol. 2020 May;17(5):541-543. doi: 10.1038/s41423-020-0401-3. Epub 2020 Mar 17. No abstract available. PMID 32203186
- [Result] Zumla A, Hui DS, Azhar EI, Memish ZA, Maeurer M. Reducing mortality from 2019-nCoV: host-directed therapies should be an option. Lancet. 2020 Feb 22;395(10224):e35-e36. doi: 10.1016/S0140-6736(20)30305-6. Epub 2020 Feb 5. No abstract available. PMID 32035018
- See also: Polymerized-Type I collagen induces a high-quality cartilage repair in a rat model of osteoarthritis — https://scidoc.org/IJBRR-2470-4520-04-201.php
- See also: Correlation Analysis Between Disease Severity and Inflammation related Parameters in Patients with COVID-19 Pneumonia — https://www.medrxiv.org/content/10.1101/2020.02.25.20025643v1
- See also: . Successful Treatment Strategy of Turkey against Covid-19 Outbreak — https://es.scribd.com/document/467773330/EDITORIAL-Successful-Treatment-Strategy-of-Turkey-against-Covid19-Outbreak-12345-pdf
- See also: Characteristics of lymphocyte subsets and cytokines in peripheral blood of 123 hospitalized patients with 2019 novel coronavirus pneumonia (NCP). — https://doi.org/10.1101/2020.02.10.20021832
- See also: Exuberant elevation of IP-10, MCP-3 and IL-1ra during SARS-CoV-2 infection is associated with disease severity and fatal outcome — https://www.medrxiv.org/content/10.1101/2020.03.02.20029975v1.full.pdf